CLINICAL TRIAL: NCT04175574
Title: Effects of Music on Pain and Anxiety During Post-operative Period in Closed Shaft Femur Fracture Patients in Serdang Hospital and University Malaya Medical Centre
Brief Title: Effects of Music on Post-operative Pain and Anxiety
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universiti Putra Malaysia (Other)
Collaborators: University of Malaya (Other)
Responsible Party: Principal Investigator, PRI CHASKAR, Postgraduate student, Universiti Putra Malaysia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: UPM2019MUSICINMEDICINE
Record Dates: First submitted 2019-09-02; First posted 2019-11-25 (Actual); Last update posted 2021-12-02 (Actual); Status verified 2021-12

CONDITIONS: Closed Fracture of Shaft of Femur; Postoperative Pain; Postoperative Anxiety
Keywords: post-operative pain relief; post-operative anxiety; non-pharmacological adjuvant; closed shaft femur fracture; randomised controlled trial
MeSH Terms: conditions — Pain, Postoperative | interventions — Music Therapy

STUDY DESIGN:
Intervention Model Description: The design of this study is a randomised controlled trial based on the CONSORT 2010 flow diagram. Patients warded at the orthopaedics wards in two government hospitals, who have been hospitalized following a closed midshaft femur fracture and planned for surgery. Patients who fulfill the inclusion criteria will be invited to participate in this study. Recruitment to participate is based on voluntary and they will be given the patient information sheet, written informed consent and briefed on the protocol of the study. The patients will be randomised either in the intervention or control group by selecting an opaque envelope.
Who Masked: Participant, Investigator
Masking Description: To ensure non-bias during the randomization, both the researcher and the patient will be masked and this procedure will be carried out by a trained research assistant.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The intervention consist of the patients in the experimental group listening to pre-recorded music played through a set of noise cancelling Sony headphones which are padded for extra comfort from a Sony Digital Walkman. The duration of the intervention is 30 minutes without interruption, such as eating, talking and being on their mobile phones.
  Interventions: Other: Music
- Control group (No Intervention): Whereas, patients in the control group will be given similar headphones but without any music. They will also be briefed not to eat, talk and being on their mobile phones.

INTERVENTIONS:
Other: Music — The music has no lyrics, has a sustained melodic quality, has no strong rhythms and percussion or base, rate of 60-80 beats per minute, promotes relaxation, calming and soothing, neutral and is unbiased towards any culture or age. The volume of the music will be pre-adjusted to the patients' preference (preferable 30 dB) by the research assistant.
  Arms: Intervention group

SUMMARY:
It has been hypothesized that because music has the ability to motivate, promote relaxation, alleviate pain and anxiety levels, to distract, and facilitate positive emotional states; thus it will enable healing by reducing anxiety levels which are associated with expected pain, hence patients are more unperturbed. In addition, several studies in the past have also identified that music listening can reduce the need for analgesics before surgery and after surgery to alleviate pain, reduce the period of post-operative pain and aid in the recovery period. While most studies which had administered music listening in the post-anaesthesia care unit (PACU), had found significant findings compared to patients that did not listen to music; there are few others which found otherwise.

Over decades, time and again, researchers have tried to understand how non-pharmacological interventions have been utilized in a spectrum of rehabilitation settings in populations to stimulate convalesces. This is because non-pharmacological interventions have been recognised as valuable, simple, safe, and inexpensive adjuvants to pharmacological approaches in pain management and therefore is valuable during post-operative rehabilitation especially.

This research is necessary because it hopes to address the gap of knowledge concerning the effects of music in post-operative pain, anxiety objectively in a specific population, and during an explicit time frame in a public hospital setting in Malaysia and whether by listening to music, the patients will require lesser amount of opioids analgesics.

The purpose of this study is to examine the effects of music on pain and anxiety during post-operative period in patients with closed shaft femur fracture at University of Malaya Medical Centre.

DETAILED DESCRIPTION:
The administration of music as an adjuvant to medicine during the recovery after surgery especially should be further explored by examining the physiological parameters of what takes place in the human body when pain and anxiety are present.

Permision to conduct this study have been granted by the National Medical Research Registry of the Ministry of Health of Malaysia, the Medical Research Ethics Committee from Universiti Putra Malaysia as well as University of Malaya.

During the intervention, the standard course of treatment by the attending physician will not be interrupted. The patients have the liberty to drop out from the study at any point of time without any repercussion.

The Standard Operating Procedure for all information obtained in this study will be kept and handled in a confidential manner, and destroyed thereafter analysis in accordance with applicable laws and regulations by the Ethics Committee of Universiti Putra Malaysia. When publishing or presenting the study results, the identity of the patients will not be revealed. Only individuals involved in this study such as the researchers, attending physicians, qualified monitors and auditors, Universiti Putra Malaysia or its affiliates and governmental or regulatory authorities can access the data from this study.

The sample size assessment to specify the number of participants was necessary to demonstrate an effect.

Data collected will be coded and transferred into the SPSS (Version 25.0) for analyses. Appropriate tests will be selected based on whether the data is normally distributed or not. P-value will be set to 0.05 to indicate level of significance with confidence interval of 95%. Depending on the distribution of the data, the appropriate statistical analysis will be determined to compare pre- and post-test results. Descriptive statistical analysis will be performed on all study variable at each time point. Spearman correlation coefficient will be used to determine the correlation of the main study outcomes, which are pain and anxiety. Inferential statistical analysis such as t-test and Chi-square will be used to determine the existence of significance differences in demography of the patients. Paired t-test will be used to differentiate the results between the pre- and post-test for the pain and anxiety scores. A normality test, Kolmogorov-Smirnov test, will be performed to look at the distribution of the data. For comparison between the experimental and control group, the Mann-Whitney U and one-way analysis of variance (ANOVA) tests will be performed to using the median and mean scores from both groups and as well the dosage of analgesia prescribed to both groups.

Missing information will be recorded but not included in the data analysis. Data collected, processed and churned for results and reported by the researcher will be closely monitored by a certified medical statistician who has been appointed to advice the research team. The supervisory committee will retain all rights to advise on the development of the research.

ELIGIBILITY:
Inclusion Criteria:

* Consent to having the surgery and general anaesthesia
* Free from cognitive impairment
* Free from non-communicable diseases
* Mentally stable
* No appreciable deficits in vision and hearing
* American Society of Anaesthesiology (ASA) physical status classification of 1, 2, or 3
* Able to communicate either in English or Bahasa Malaysia
* Admitted to the Orthopaedic ward post-operatively
* Alert and cognizant to complete the pain and anxiety scores

Exclusion Criteria:

* Patient refusal for surgery and anaesthesia
* Patients anticipated to have difficult airway and planned for higher level airway management such as awake fibreoptic intubation, tracheostomy under local anaesthetic.
* Patients who are cognitively impaired
* Women under hormonal treatment
* Diagnosed with auto immune disease
* Deaf and vision impaired
* Current use of anti-psychotic medication
* Haemodynamically not stable

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 108 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Pain score using the Numeric Rating Scale (NRS) | The change between the baseline and post-intervention will be assessed. The intervention is for 30 minutes long and will be administered 24 hours post surgery.
  Mean score of pain level (1-3 = mild; 4-6 = moderate; 7-10 = severe)
Brief Pain Inventory (BPI) | The change between the baseline and post-intervention will be assessed. The intervention is for 30 minutes long and will be administered 24 hours post surgery.
  Worst, least and average pain in the last 24 hours
Anxiety score using the Generalized Anxiety Disorder-7 (GAD-7) | The change between the baseline and post-intervention will be assessed. The intervention is for 30 minutes long and will be administered 24 hours post surgery.
  Mean score of anxiety level (0-4 = minimal anxiety; 5-9 = mild anxiety; 10-14 = moderate anxiety; 15-21 severe anxiety)

SECONDARY OUTCOMES:
Opioid dosage | 48 hours post surgery
  Average amount of opioids (mg) ingested between the intervention and control group
Pro-inflammatory cytokine Interleukin 6 (IL-6) | The change between the baseline and post-intervention will be assessed. The intervention is for 30 minutes long and will be administered 24 hours post surgery
  Pro-inflammatory cytokine Interleukin 6 (IL-6) (pg)
Cortisol level | The change between the baseline and post-intervention will be assessed. The intervention is for 30 minutes long and will be administered 24 hours post surgery
  Cortisol level (microlitres)
Heart Rate | The change between the baseline and post-intervention will be assessed. The intervention is for 30 minutes long and will be administered 24 hours post surgery
  Heart rate (bpm)
Respiratory Rate | The change between the baseline and post-intervention will be assessed. The intervention is for 30 minutes long and will be administered 24 hours post surgery
  Respiratory rate (breaths per minute)
Systolic and diastolic Blood pressure | The change between the baseline and post-intervention will be assessed. The intervention is for 30 minutes long and will be administered 24 hours post surgery
  Systolic and diastolic Blood pressure (mmHg)
Oxygen saturation | The change between the baseline and post-intervention will be assessed. The intervention is for 30 minutes long and will be administered 24 hours post surgery
  Oxygen saturation (%)

CONTACTS AND LOCATIONS:
Locations (1):
- Serdang Hospital, Serdang, Selangor, Malaysia

IPD SHARING:
Plan to Share IPD: No